CLINICAL TRIAL: NCT02705352
Title: A Prospective, Randomized, Double-blinded Comparison of the Use of 5-fluorouracil Versus Placebo in Periocular Full Thickness Skin Grafts.
Brief Title: 5-fluorouracil Versus Placebo in Periocular Full Thickness Skin Grafts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Michael Yoon, Ophthalmic Plastic and Reconstructive Surgery Attending, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 786680-1
Record Dates: First submitted 2016-02-22; First posted 2016-03-10 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Ectropion; Skin Neoplasms
Keywords: Skin graft; 5-Fluorouracil; Periocular reconstruction
MeSH Terms: conditions — Ectropion; Skin Neoplasms | interventions — Fluorouracil; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-Fluorouracil (Experimental): Antimetabolite will be injected 2 weeks after periocular reconstruction with full thickness skin graft. Injection will be repeated every 2 weeks for a total of up to 4 injections.
  Interventions: Drug: 5-Fluorouracil
- Normal saline (Placebo Comparator): Normal saline will be injected 2 weeks after periocular reconstruction with full thickness skin graft. Injection will be repeated every 2 weeks for a total of up to 4 injections.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: 5-Fluorouracil — Treatment medication
  Other Names: 5-FU
  Arms: 5-Fluorouracil
Other: Normal saline — Placebo
  Other Names: Saline
  Arms: Normal saline

SUMMARY:
Full thickness skin grafts are an essential tool in surgery around the eyelids for reconstruction or rehabilitation following injury or surgery. Common conditions where skin grafts are needed include cicatricial ectropion, restoration of eyelid function after tumor removal, burns to the eyelids, or trauma. Early complications, occurring in the first 2 weeks after surgery, are rare: wound dehiscence, necrosis, infection, bleeding, partial or complete graft failure. However, late postoperative complications generally categorized as "scarring" (including graft hypertrophy and contraction, keloid formation, and hypo/hyper pigmentation) can limit the success and acceptability of the procedure by patients. Scars form following any insult to the deep dermis as a result of wound healing. Factors such as age, skin type, racial pigmentation, genetics, and sex may influence fibroblast proliferation as part of the healing response, resulting in a suboptimal result. Graft contraction is perhaps the most worrisome result, since it can result in failure of the initial surgery and may require additional surgery to correct. Many treatments have been used to manage these complications: corticosteroid injection, cryotherapy, pressure therapy, radiotherapy, laser therapy, silicone based products, and antimetabolite therapy. One such antimetabolite, 5-fluorouracil (5-FU), has been used over the last 15 years as an adjunct or primary treatment to modulate wound healing and scar formation. Other studies have demonstrated safety for cutaneous and subcutaneous injection in the periocular region. However, no controlled studies exist. This prospective, randomized, and double-blinded clinical study will evaluate the use and benefit of 5-FU versus saline in patients undergoing skin grafting for periocular reconstruction. The decision for the need for skin grafting will be at the discretion of the attending surgeon and will be made separate from enrollment in the study. Surgery will be performed as indicated. The study medication or placebo (normal saline) will be administered 2-3 weeks after surgery and then every 2-3 weeks afterwards for up to a total of 4 injections. After the injections, regular scheduled follow-up will be at 3, 6, and 12 months post-op. Outcomes at each study visit (up to 12 months post-operatively) include graft size, color, contour, and complications between study treatment group and placebo group.

DETAILED DESCRIPTION:
In oculofacial surgery, full thickness skin grafts are a fundamental tool used to restore function to the eyelid. This can be required after removal of skin cancer, correction of eyelid malposition such as cicatricial eyelid ectropion (the eyelid edge is pulled away from the eye), retraction (the eyelid is pulled lower than normal, exposing more of the eye to the air), scar formation (such as a medial pulling or web), or trauma with loss of tissue. These conditions affect patients of all ages, ranging from newborns to nonagenarians. Skin grafting in the periorbital area is relatively safe, although complications may arise. The most common and challenging complication scarring and graft shrinkage. This can lead to requiring additional surgery to add additional skin or to improve the appearance of the graft. In addition to the morbidity of another surgery, some patients have limited or no additional skin available (e.g. young patients, burn patients). The eyelid skin is the thinnest of the body, so only thin skin can be used as donor material. However, the amount of skin available for this purpose is very little.

There are limited options for preventing graft shrinkage and scarring in this situation. The oldest and most commonly used technique is injection of steroid medication. Steroids decrease proliferation of a fibroblast cells, which create collagen and glycosaminoglycan, two proteins created by the body that contract and cause graft shrinkage. Data in literature shows that one form of steroid, triamcinolone, is effective for this purpose. However, there is a risk of embolization of this solid steroid material that care rarely cause blindness. In addition, in the periocular area, steroids can elevate eye (intraocular) pressure (that can cause glaucoma in some cases) and accelerate the formation of cataracts.

Another medication used for this purpose is 5-fluorouracil (5-FU). This is an antimetabolite (a drug that inhibits another chemical that is part of normal processes) that works by irreversibly inhibiting the enzyme thymidylate synthetase resulting in impaired DNA synthesis. This reduces fibroblast proliferation and inhibits collagen type 1 production which is a key protein in scar formation. This medication is commonly used in ophthalmology after glaucoma filtration surgery. In this usage, it is injected under the conjunctiva to prevent scarring around the surgical site.

There have been two retrospective studies that have investigated the safety and efficacy of 5-FU injected in periorbital skin grafts with or without Kenalog. The first (Massry 2011) used post-operative injections of a 50:50 mixture of 5-FU and triamcinolone for correction of medial canthal webs. In 2 patients, they found it to be safe and effective. The author noted he has used it previously for other scar management cases and was "very pleased with the results and [had] negligible side-effect[s]." The same author performed another study using 5-FU for skin grafts. This study evaluated 19 patients who had skin grafts for various purposes and were injected following surgery (similar to our protocol). This study demonstrated safety of the injection, with no cases of complication. The author concluded that the 5-FU is effective with "minimal scarring, high patient and surgeon satisfaction, and few complications." However, there was no comparison group to truly evaluate the effect. With only two retrospective studies by the same author, there is no strong evidence that it is effective, although safety has been demonstrated.

The investigators therefore propose a randomized controlled prospective study to evaluate the outcomes of periocular skin grafts with or without the use of 5-FU injected in the post-operative period. Patients will be recruited from the investigators' practices who need full thickness skin grafts for reconstruction after cancer removal, pre-existing scarring, eyelid malposition, or trauma. Patients will be introduced to the study, and will come back for detailed explanation and consent. The injection medication will be prepared by the Mass Eye and Ear Research Pharmacy and labeled for this double-blinded study. Injections will be given 2-3 weeks after surgery and up to 4 times (also every 2-3 weeks). Measurements and photographs of the skin graft will be taken at each visit (following injections, at 3, 6, and 12 months) to monitor for complications. Patients will be followed for at least 12 months.

If effective, this medication could change the post-operative management of skin grafts, reduce complications and reoperations.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Ages 18 to 89 years of age
* Has a condition (e.g. trauma, skin/tissue defect, scar) requiring a skin graft for repair
* Sufficient education to understand study procedures and to give consent

Exclusion Criteria:

* Women lactating, pregnant or planning to get pregnant in the near future
* Immunosuppression/immunocompromise or serious/active infections
* Dihydropyrimidine dehydrogenase enzyme deficiency
* Severe hepatic or renal impairment or failure
* Unable to give consent or understand the study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-08-25 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Yoon, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Challenges recruiting patients into the study.
Period: Overall Study
Arm/Group | 5-Fluorouracil | Normal Saline
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Unable to recruit patients into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | 5-Fluorouracil | Normal Saline | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 1 |  | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (0) |  | 72 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1
Scar appearance [Number; unit: units on a scale] — Patient and Observer Scar Assessment Scale (POSAS). This has 2 parts: Patient and Observer Scale. Both contain 6 items scored numerically on a 10 step scale (1 most normal, 10 worst scar imaginable). Together they sum to 'Total Score' of the Patient and Observer Scale. Category boxes are available to score nominal parameters (e.g. type of colour). Moreover, the patient and observer also score their 'Overall Opinion'. Total and subscales are averaged.
  *There was 1 participant, and the score average was 1.*
  units on a scale | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Graft Size Change
Description: Full thickness skin grafts will be measured prior to treatment (at time of surgery) and 12 months after surgery. Although the graft will be measured at each visit, the outcome is the percent change from baseline at 12 months.
Time Frame: 12 months
Population: One white male in study group
Measure: Number; unit: percent change in graft
Arm/Group | 5-Fluorouracil | Normal Saline
Number analyzed (Participants) | 1 | 0
percent change in graft | 10 |

2. Secondary Outcome: Adverse Events
Description: Treatment side effects will be recorded. Examples include pain, skin thinning, color/texture change, atrophy, telangiectasis, infection, and erythema.
Time Frame: 12 months
Population: Unable to recruit more study patients.
Measure: Number; unit: Events
Arm/Group | 5-Fluorouracil | Normal Saline
Number analyzed (Participants) | 1 | 0
Events | 0 |

3. Secondary Outcome: Early Post-operative Complications
Description: Surgery complications will be recorded, not related to treatment. Examples are wound dehiscence, graft necrosis, infection, bleeding, partial/complete graft failure and/or ectropion.
Time Frame: 2 weeks after surgery
Population: Unable to recruit more study patients.
Measure: Number; unit: Number of events
Arm/Group | 5-Fluorouracil | Normal Saline
Number analyzed (Participants) | 1 | 0
Number of events | 0 |

4. Secondary Outcome: Surgeon and Patient Satisfaction
Description: Patient and Observer Scar Assessment Scale (POSAS). This has 2 parts: Patient and Observer Scale. Both contain 6 items scored numerically on a 10 step scale (1 most normal, 10 worst scar imaginable). Together they sum to 'Total Score' of the Patient and Observer Scale. Category boxes are available to score nominal parameters (e.g. type of colour). Moreover, the patient and observer also score their 'Overall Opinion'. Total and subscales are averaged.
  *There was 1 participant, and the score average was 1.*
Time Frame: 12 months
Population: Unable to recruit more patients.
Measure: Number; unit: score on a scale
Arm/Group | 5-Fluorouracil | Normal Saline
Number analyzed (Participants) | 1 | 0
score on a scale | 1 |

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | 5-Fluorouracil | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT02705352/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT02705352/SAP_001.pdf